CLINICAL TRIAL: NCT05011110
Title: Prospective Assessment to Evaluate the Ease of Application and Removal of GraduSOX™ VLU Kit Compared to Sigvaris™ Ulcer X VLU Kit, and Comfort in Use by Healthy Patients Who Have Completed Venous Treatment
Brief Title: Evaluating the Ease of Application, Removal, and Comfort of Gradusox™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Whiteley Clinic (Other)
Collaborators: VeinSense (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TWC-AC-2021-01
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Ease of Applying and Removing, and Comfort, of Compression Stockings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GraduSOX (left leg) & Sigvaris (right leg) (Experimental): Half of participants will wear a GraduSOX compression stocking on their left leg whilst wearing a Sigvaris compression stocking on their right leg.
  Interventions: Device: Graduated compression stockings
- GraduSOX (right leg) & Sigvaris (left leg) (Experimental): Half of participants will wear a GraduSOX compression stocking on their right leg whilst wearing a Sigvaris compression stocking on their left leg.
  Interventions: Device: Graduated compression stockings

INTERVENTIONS:
Device: Graduated compression stockings — Both GraduSOX and Sigvaris are graduated compression stockings. These exert the greatest degree of of compression at the ankle, and the level of compression gradually decreases up the garment.
  Other Names: GraduSOX; Sigvaris

SUMMARY:
The aims of this study are to evaluate the comfort, and ease of application and removal, of GraduSOX™ compression stockings compared to standard compression stockings of the same compression class.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will be randomised by closed envelope randomisation to either a) GraduSOX on their right leg and Sigvaris on their left leg, or b) Sigvaris on their right leg and GraduSOX on their left leg. At Day 1, participants will attend the clinic and be fitted with their stockings and given an Evaluation Form. The Evaluation Form has four sections to be completed on Day 1, Day 2, Day 4 and Day 8 of the study. Each section asks multiple choice questions related to the comfort and ease of applying and removing each stocking.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over.
* Have known previous venous insufficiency that has been treated.
* Have no known current contraindication to the wearing of graduated compression hosiery.
* Have an ankle brachial pressure index (ABPI) between 0.8-1.2.
* Have no active ulceration.
* Are physically able to apply and remove hosiery kits safely.
* Have had successful surgery at The Whiteley Clinic and have had at least one follow-up to show no residual venous disease.

Exclusion Criteria:

* Under the age of 18.
* Have known arterial insufficiency (an ABPI of below 0.8).
* Have active ulceration.
* Be physically unable to put stocking on their own legs.
* Have signs of recent lower limb trauma, active infection, ongoing untreated venous disease, significant ankle oedema.
* Unable to give informed consent.
* Pregnant.
* Fragile skin that may be damaged whilst trying to apply or remove compression stockings.
* Previous DVT or complicated varicose veins that were not able to be completely treated and left residual venous reflux disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that graded Gradusox stockings as easier to apply compared to Sigvaris. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to apply compared to Gradusox. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as easier to remove compared to Sigvaris. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to remove compared to Gradusox. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as more comfortable compared to Sigvaris. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Sigvaris stockings as more comfortable compared to Gradusox. | Day 1 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Gradusox stockings as easier to apply compared to Sigvaris. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to apply compared to Gradusox. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as easier to remove compared to Sigvaris. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to remove compared to Gradusox. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as more comfortable compared to Sigvaris. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Sigvaris stockings as more comfortable compared to Gradusox. | Day 2 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Gradusox stockings as easier to apply compared to Sigvaris. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to apply compared to Gradusox. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as easier to remove compared to Sigvaris. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to remove compared to Gradusox. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as more comfortable compared to Sigvaris. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Sigvaris stockings as more comfortable compared to Gradusox. | Day 4 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Gradusox stockings as easier to apply compared to Sigvaris. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to apply compared to Gradusox. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as easier to remove compared to Sigvaris. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Sigvaris stockings as easier to remove compared to Gradusox. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very easy', 2 is 'fairly easy', 3 is 'neither easy nor difficult', 4 is 'quite difficult', and 5 is 'very difficult'.
Number of participants that graded Gradusox stockings as more comfortable compared to Sigvaris. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.
Number of participants that graded Sigvaris stockings as more comfortable compared to Gradusox. | Day 8 of 8
  Participants use a 5-point discrete linear analogue scale 1-5, where 1 is 'very comfortable', 2 is 'comfortable', 3 is 'neither comfortable nor uncomfortable', 4 is 'uncomfortable', and 5 is 'very uncomfortable'.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS FRCS(Gen) MBBS, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants that are enrolled in the study will be assigned a unique Trial ID which will be used to anonymise the data they provide on the Evaluation Form.

REFERENCES:
- [Background] Briggs M, Flemming K. Living with leg ulceration: a synthesis of qualitative research. J Adv Nurs. 2007 Aug;59(4):319-28. doi: 10.1111/j.1365-2648.2007.04348.x. Epub 2007 Jul 2. PMID 17608682
- [Background] Ashby RL, Gabe R, Ali S, Adderley U, Bland JM, Cullum NA, Dumville JC, Iglesias CP, Kang'ombe AR, Soares MO, Stubbs NC, Torgerson DJ. Clinical and cost-effectiveness of compression hosiery versus compression bandages in treatment of venous leg ulcers (Venous leg Ulcer Study IV, VenUS IV): a randomised controlled trial. Lancet. 2014 Mar 8;383(9920):871-9. doi: 10.1016/S0140-6736(13)62368-5. Epub 2013 Dec 6. PMID 24315520
- [Background] Raju S, Hollis K, Neglen P. Use of compression stockings in chronic venous disease: patient compliance and efficacy. Ann Vasc Surg. 2007 Nov;21(6):790-5. doi: 10.1016/j.avsg.2007.07.014. PMID 17980798
- [Background] O'Meara S, Cullum N, Nelson EA, Dumville JC. Compression for venous leg ulcers. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD000265. doi: 10.1002/14651858.CD000265.pub3. PMID 23152202
- See also: Power (sample size) calculator — https://www.sealedenvelope.com/power/continuous-superiority/